CLINICAL TRIAL: NCT00732524
Title: Combination of Sulfonylureas and Insulin Glargine as Safety Net Outpatient Therapy for Unstable Diabetes and Impending Diabetic Ketoacidosis (DKA)
Brief Title: Combination of Sulfonylureas and Insulin Glargine Outpatient Therapy for Unstable Diabetes and Impending DKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Dr. Leon Fogelfeld, John H. Stroger Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #04-128
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Type 2 Diabetes
Keywords: Hyperglycemia; Glucose toxicity; Glargine; Glipizide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Glipizide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glipizide arm (Active Comparator): Glipizide XL is an insulin secretagogue and is an extended release tablet designed to provide a controlled rate of delivery. Glipizide XL was chosen because it is the most frequently used discharge oral medication in our ED. It has a quick onset of action within a few hours after oral ingestion, lasts for 24 hours and has a powerful glucose lowering effect. In addition, there are very few contraindications to Glipizide XL and there is published literature regarding their use in subjects with severe hyperglycemia
  Interventions: Drug: Glipizide
- Glipizide + Glargine (Active Comparator): Insulin Glargine is a recombinant human basal insulin analog. It was chosen since it is a non-peaking insulin with cover for 24 hours. It can be injected subcutaneously only once a day and has a low incidence of hypoglycemia
  Interventions: Drug: Glipizide and Glargine

INTERVENTIONS:
Drug: Glipizide — Glipizide XL 10 mg once daily 30 mins before breakfast
  Other Names: Glucotrol XL
  Arms: Glipizide arm
Drug: Glipizide and Glargine — Glipizide XL 10 mg daily 30 minutes before breakfast Insulin Glargine 10 units subcutaneously at bedtime daily
  Other Names: Insulin Lantus
  Arms: Glipizide + Glargine

SUMMARY:
The purpose of this study is to compare two simple and safe emergency department discharge therapy for Type 2 Diabetes patients with severe hyperglycemia and with no indications for inpatient admission.

DETAILED DESCRIPTION:
This study is an open label randomized controlled trial in adult DM2 patients seen in ED services at John H. Stroger Hospital of Cook County serving a largely uninsured/underserved population. Individuals more than 18 years of age with DM2, either with new onset DM2 or known diabetics who did not take oral hypoglycemic agents for more than 2 weeks, presenting with fasting blood glucose (FBG) 300-500 mg/dl or random blood glucose (RBG) 400-700 mg/dl and who did not have any exclusion criteria listed in Table 1, were eligible for the study. Subjects were randomized to one of the two fixed dose treatment groups: 1) Glipizide XL 10 mg orally daily prior to breakfast (G group), 2) Glipizide XL 10 mg orally daily along with Insulin Glargine 10 units at bedtime, subcutaneously (G+G group).

ELIGIBILITY:
Inclusion Criteria:

* Individuals more than 18 years of age with DM2, either with new onset DM2 or known diabetics who did not take oral hypoglycemic agents for more than 2 weeks, presenting with fasting blood glucose (FBG) 300-500 mg/dl or random blood glucose (RBG) 400-700 mg/dl and who did not have any exclusion criteria listed in Table 1, were eligible for the study.

Exclusion Criteria:

* Acute metabolic complications (diabetic ketoacidosis, hyperosmolar hyperglycemia associated with dehydration).
* Acute complications of chronic cardiovascular, neurological, renal, and other diabetic complications.
* Any subject with unstable vitals signs (temperature > 101 degrees F, systolic blood pressure < 90 or > 180 mm hg, diastolic blood pressure < 60 or > 110 mm hg, heart rate < 60 or > 120 beats/minute).
* Electrolyte imbalances (serum bicarbonate level < 20 mEq/L, serum sodium < 125 & > 150 mEq/L, serum potassium < 3.5 & > 5.5 mEq/L).
* Evidence of an impaired sensorium and/or dementia.
* Age > 75 years
* Subjects with any acute medical illness.
* Type 1 diabetes or type 2 diabetics weighing less than 120 lbs
* Current addiction to illicit substances or alcohol abuse
* Pregnant or lactating subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the patients' ability to avoid repeat ED visits or hospitalization in either of the discharge regimens. | 2 months

SECONDARY OUTCOMES:
The secondary outcomes included the number of subjects who reached a fasting or pre-meal BG goal of 80 to 130 mg/dl and assessment of the beta cell function at the beginning and end of the study as measured by C-peptide levels during OGTT testing. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Leon A Fogelfeld, MD, Principal Investigator — John H Stroger Hospital Of Cook County
Locations (1):
- John H Stroger Hospital Of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Background] Davidson MB. Successful treatment of markedly symptomatic patients with type II diabetes mellitus using high doses of sulfonylurea agents. West J Med. 1992 Aug;157(2):199-200. No abstract available. PMID 1441492
- [Background] Gleason CE, Gonzalez M, Harmon JS, Robertson RP. Determinants of glucose toxicity and its reversibility in the pancreatic islet beta-cell line, HIT-T15. Am J Physiol Endocrinol Metab. 2000 Nov;279(5):E997-1002. doi: 10.1152/ajpendo.2000.279.5.E997. PMID 11052953
- [Background] Peters AL, Davidson MB. Maximal dose glyburide therapy in markedly symptomatic patients with type 2 diabetes: a new use for an old friend. J Clin Endocrinol Metab. 1996 Jul;81(7):2423-7. doi: 10.1210/jcem.81.7.8675555.